CLINICAL TRIAL: NCT00790335
Title: Acute Venous Thrombosis: Thrombus Removal With Adjunctive Catheter-Directed Thrombolysis--The ATTRACT Trial
Brief Title: Acute Venous Thrombosis: Thrombus Removal With Adjunctive Catheter-Directed Thrombolysis
Acronym: ATTRACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: McMaster University (Other); Ontario Clinical Oncology Group (OCOG) (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); BSN Medical Inc (Industry); Genentech, Inc. (Industry); Medtronic - MITG (Industry); Boston Scientific Corporation (Industry); Mid America Heart Institute (Other); Society of Interventional Radiology Foundation (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22326953211; U01HL088476-01A1 (NIH)
Record Dates: First submitted 2008-10-15; First posted 2008-11-13 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Deep Vein Thrombosis; Venous Thrombosis; Postphlebitic Syndrome; Venous Thromboembolism; Post Thrombotic Syndrome
Keywords: deep vein thrombosis; deep venous thrombosis; post thrombotic syndrome; blood clot; thrombolysis; tissue plasminogen activator; rt-PA; Activase; mechanical thrombectomy; pharmacomechanical; ATTRACT
MeSH Terms: conditions — Venous Thrombosis; Postphlebitic Syndrome; Venous Thromboembolism; Postthrombotic Syndrome; Thrombosis | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-Intervention (Experimental): PCDT with intrathrombus delivery of recombinant tissue plasminogen activator (rt-PA, maximum allowable total dose 35 mg) into the DVT over a period of up to 24 hours. Three methods of initial rt-PA delivery will be used: 1) Trellis-8 Peripheral Infusion System - maximum first-session rt-PA dose 25 mg; 2) AngioJet Rheolytic Thrombectomy System - maximum first-session rt-PA dose 25 mg; or 3) Catheter-directed rt-PA infusion for up to 24 hours at 0.01 mg/kg/hr (maximum 1.0 mg/hr) via a multisidehole infusion catheter. Before and after PCDT, patients will receive standard DVT therapy as in the Control Arm
  Interventions: Drug: Recombinant tissue plasminogen activator (rt-PA)
- B-Control (No Intervention): Initial anticoagulant therapy with unfractionated heparin, enoxaparin, dalteparin, or tinzaparin, for at least 5 days, overlapped with long-term oral warfarin (target international normalized ratio 2.0 - 3.0). Elastic compression stockings will be prescribed

INTERVENTIONS:
Drug: Recombinant tissue plasminogen activator (rt-PA) — Pharmacomechanical catheter-directed thrombolysis, consisting of intrathrombus administration of rt-PA using a catheter/device.
  Other Names: rt-PA; recombinant tissue plasminogen activator; Activase; Alteplase
  Arms: A-Intervention

SUMMARY:
The purpose of this study is to determine if the use of adjunctive Pharmacomechanical Catheter Directed Thrombolysis, which includes the intrathrombus administration of rt-PA--Activase (Alteplase),can prevent the post-thrombotic syndrome(PTS)in patients with symptomatic proximal deep vein thrombosis(DVT)as compared with optimal standard DVT therapy alone.

DETAILED DESCRIPTION:
Activase, the study drug, is a fibrinolytic drug that is indicated for use in acute myocardial infarction, acute ischemic stroke, and acute massive pulmonary embolism in adults. Previous studies have established the ability of rt-PA to lyse venous thrombus in patients with deep vein thrombosis (DVT), and suggest that successful rt-PA mediated thrombolysis can prevent the post-thrombotic syndrome (PTS), a morbid, late complication of DVT that occurs in nearly 50% of patients.

rt-PA is delivered directly into venous thrombus using a catheter/device which is embedded within the thrombus by a physician under imaging guidance. This method of rt-PA delivery, pharmacomechanical catheter-directed intrathrombus thrombolysis (PCDT),is thought to be safer, more effective, and more efficient than previous methods. The question of whether PCDT using rt-PA improves long-term DVT patient outcomes with acceptable risk and cost has not yet been addressed.

The rationale for performing the ATTRACT Trial is based upon:

* the major burden of PTS on DVT patients and the U.S. healthcare system
* the association between rapid clot lysis and prevention of PTS
* the proven ability of rt-PA to dissolve venous thrombus in proximal DVT
* recent advances in CDT methods which may lower bleeding risk
* the major clinical controversy on whether CDT should be routinely used for first-line DVT therapy

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic proximal DVT involving the iliac, common femoral, and/or femoral vein.

Exclusion Criteria:

* Age less than 16 years or greater than 75 years.
* Symptom duration > 14 days for the DVT episode in the index leg (i.e., non-acute DVT).
* In the index leg: established PTS, or previous symptomatic DVT within the last 2 years.
* In the contralateral (non-index) leg: symptomatic acute DVT a) involving the iliac and/or common femoral vein; or b) for which thrombolysis is planned as part of the initial therapy.
* Limb-threatening circulatory compromise.
* Pulmonary embolism with hemodynamic compromise (i.e., hypotension).
* Inability to tolerate PCDT procedure due to severe dyspnea or acute systemic illness.
* Allergy, hypersensitivity, or thrombocytopenia from heparin, rt-PA, or iodinated contrast, except for mild-moderate contrast allergies for which steroid pre-medication can be used.
* Hemoglobin < 9.0 mg/dl, INR > 1.6 before warfarin was started, or platelets < 100,000/ml.
* Moderate renal impairment in diabetic patients (estimated glomerular filtration rate [GFR] < 60 ml/min) or severe renal impairment in non-diabetic patients (estimated GFR < 30 ml/min).
* Active bleeding, recent (< 3 mo) GI bleeding, severe liver dysfunction, bleeding diathesis.
* Recent (< 3 mo) internal eye surgery or hemorrhagic retinopathy; recent (< 10 days) major surgery, cataract surgery, trauma, cardiopulmonary resuscitation, obstetrical delivery, or other invasive procedure.
* History of stroke or intracranial/intraspinal bleed, tumor, vascular malformation, aneurysm.
* Active cancer (metastatic, progressive, or treated within the last 6 months). Exception: patients with non-melanoma primary skin cancers are eligible to participate in the study.
* Severe hypertension on repeated readings (systolic > 180 mmHg or diastolic > 105 mmHg).
* Pregnant (positive pregnancy test, women of childbearing potential must be tested).
* Recently (< 1 mo) had thrombolysis or is participating in another investigational drug study.
* Use of a thienopyridine antiplatelet drug (except clopidogrel) in the last 5 days.
* Life expectancy < 2 years or chronic non-ambulatory status.
* Inability to provide informed consent or to comply with study assessments (e.g. due to cognitive impairment or geographic distance).

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2009-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Vedantham, M.D., Principal Investigator — Clinical Coordinating Center at Washington University School of Medicine; Clive Kearon, MB, MRCP, FRCP(C), PhD, Principal Investigator — Data Coordinating Center at McMaster University-Ontario Clinical Oncology Group; Samuel Z Goldhaber, M.D., Study Chair — Brigham and Women's Hospital
Locations (56):
- United States (56):
  - Arrowhead Hospital/Phoenix Heart, PLLC, Glendale, Arizona
  - St. Joseph Hospital, Orange, California
  - Stanford University Medical Center, Stanford, California
  - Danbury Hospital, Danbury, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Christiana Care Health Systems, Newark, Delaware
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Mease Countryside Hospital, Clearwater, Florida
  - Baptist Cardiac & Vascular Institute, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Florida Hospital-Tampa Division-Pepin Heart Institute and Dr. Kiran C. Patel Research Institute, Tampa, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Adventist Midwest Health, Hinsdale, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - CorVasc, Indianapolis, Indiana
  - University of Iowa Carver's College of Medicine, Iowa City, Iowa
  - St. Elizabeth Healthcare of Northern Kentucky, Florence, Kentucky
  - Maine Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ann Arbor Veteran's Administration Health System, Ann Arbor, Michigan
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Holy Name Hospital, Teaneck, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Cornell Weill Medical Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Jobst Vascular Center, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - The Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Utah Valley Regional Medical Center, Provo, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Sacred Heart Medical Center, Spokane, Washington
  - Gundersen Clinic, Ltd., La Crosse, Wisconsin
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Background] Kearon C, Kahn SR, Agnelli G, Goldhaber S, Raskob GE, Comerota AJ. Antithrombotic therapy for venous thromboembolic disease: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):454S-545S. doi: 10.1378/chest.08-0658. PMID 18574272
- [Background] Kahn SR. The post-thrombotic syndrome: the forgotten morbidity of deep venous thrombosis. J Thromb Thrombolysis. 2006 Feb;21(1):41-8. doi: 10.1007/s11239-006-5574-9. PMID 16475040
- [Background] Vedantham S, Millward SF, Cardella JF, Hofmann LV, Razavi MK, Grassi CJ, Sacks D, Kinney TB; Society of Interventional Radiology. Society of Interventional Radiology position statement: treatment of acute iliofemoral deep vein thrombosis with use of adjunctive catheter-directed intrathrombus thrombolysis. J Vasc Interv Radiol. 2006 Apr;17(4):613-6. doi: 10.1097/01.RVI.0000203802.35689.66. No abstract available. PMID 16614142
- [Background] Vedantham S, Vesely TM, Sicard GA, Brown D, Rubin B, Sanchez LA, Parti N, Picus D. Pharmacomechanical thrombolysis and early stent placement for iliofemoral deep vein thrombosis. J Vasc Interv Radiol. 2004 Jun;15(6):565-74. doi: 10.1097/01.rvi.0000127894.00553.02. PMID 15178716
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829
- [Derived] Li W, Kessinger CW, Orii M, Lee H, Wang L, Weinberg I, Jaff MR, Reed GL, Libby P, Tawakol A, Henke PK, Jaffer FA. Time-Restricted Salutary Effects of Blood Flow Restoration on Venous Thrombosis and Vein Wall Injury in Mouse and Human Subjects. Circulation. 2021 Mar 23;143(12):1224-1238. doi: 10.1161/CIRCULATIONAHA.120.049096. Epub 2021 Jan 15. PMID 33445952
- [Derived] Kahn SR, Julian JA, Kearon C, Gu CS, Cohen DJ, Magnuson EA, Comerota AJ, Goldhaber SZ, Jaff MR, Razavi MK, Kindzelski AL, Schneider JR, Kim P, Chaer R, Sista AK, McLafferty RB, Kaufman JA, Wible BC, Blinder M, Vedantham S; ATTRACT Trial Investigators. Quality of life after pharmacomechanical catheter-directed thrombolysis for proximal deep venous thrombosis. J Vasc Surg Venous Lymphat Disord. 2020 Jan;8(1):8-23.e18. doi: 10.1016/j.jvsv.2019.03.023. PMID 31843251
- [Derived] Magnuson EA, Chinnakondepalli K, Vilain K, Kearon C, Julian JA, Kahn SR, Goldhaber SZ, Jaff MR, Kindzelski AL, Herman K, Brady PS, Sharma K, Black CM, Vedantham S, Cohen DJ. Cost-Effectiveness of Pharmacomechanical Catheter-Directed Thrombolysis Versus Standard Anticoagulation in Patients With Proximal Deep Vein Thrombosis: Results From the ATTRACT Trial. Circ Cardiovasc Qual Outcomes. 2019 Oct;12(10):e005659. doi: 10.1161/CIRCOUTCOMES.119.005659. Epub 2019 Oct 8. PMID 31592728
- [Derived] Weinberg I, Vedantham S, Salter A, Hadley G, Al-Hammadi N, Kearon C, Julian JA, Razavi MK, Gornik HL, Goldhaber SZ, Comerota AJ, Kindzelski AL, Schainfeld RM, Angle JF, Misra S, Schor JA, Hurst D, Jaff MR; ATTRACT Trial Investigators. Relationships between the use of pharmacomechanical catheter-directed thrombolysis, sonographic findings, and clinical outcomes in patients with acute proximal DVT: Results from the ATTRACT Multicenter Randomized Trial. Vasc Med. 2019 Oct;24(5):442-451. doi: 10.1177/1358863X19862043. Epub 2019 Jul 27. PMID 31354089
- [Derived] Kearon C, Gu CS, Julian JA, Goldhaber SZ, Comerota AJ, Gornik HL, Murphy TP, Lewis L, Kahn SR, Kindzelski AL, Slater D, Geary R, Winokur R, Natarajan K, Dietzek A, Leung DA, Kim S, Vedantham S. Pharmacomechanical Catheter-Directed Thrombolysis in Acute Femoral-Popliteal Deep Vein Thrombosis: Analysis from a Stratified Randomized Trial. Thromb Haemost. 2019 Apr;119(4):633-644. doi: 10.1055/s-0039-1677795. Epub 2019 Jan 30. PMID 30699446
- [Derived] Comerota AJ, Kearon C, Gu CS, Julian JA, Goldhaber SZ, Kahn SR, Jaff MR, Razavi MK, Kindzelski AL, Bashir R, Patel P, Sharafuddin M, Sichlau MJ, Saad WE, Assi Z, Hofmann LV, Kennedy M, Vedantham S; ATTRACT Trial Investigators. Endovascular Thrombus Removal for Acute Iliofemoral Deep Vein Thrombosis. Circulation. 2019 Feb 26;139(9):1162-1173. doi: 10.1161/CIRCULATIONAHA.118.037425. PMID 30586751
- [Derived] Vedantham S, Goldhaber SZ, Julian JA, Kahn SR, Jaff MR, Cohen DJ, Magnuson E, Razavi MK, Comerota AJ, Gornik HL, Murphy TP, Lewis L, Duncan JR, Nieters P, Derfler MC, Filion M, Gu CS, Kee S, Schneider J, Saad N, Blinder M, Moll S, Sacks D, Lin J, Rundback J, Garcia M, Razdan R, VanderWoude E, Marques V, Kearon C; ATTRACT Trial Investigators. Pharmacomechanical Catheter-Directed Thrombolysis for Deep-Vein Thrombosis. N Engl J Med. 2017 Dec 7;377(23):2240-2252. doi: 10.1056/NEJMoa1615066. PMID 29211671
- [Derived] Vedantham S, Goldhaber SZ, Kahn SR, Julian J, Magnuson E, Jaff MR, Murphy TP, Cohen DJ, Comerota AJ, Gornik HL, Razavi MK, Lewis L, Kearon C. Rationale and design of the ATTRACT Study: a multicenter randomized trial to evaluate pharmacomechanical catheter-directed thrombolysis for the prevention of postthrombotic syndrome in patients with proximal deep vein thrombosis. Am Heart J. 2013 Apr;165(4):523-530.e3. doi: 10.1016/j.ahj.2013.01.024. Epub 2013 Mar 5. PMID 23537968
- [Derived] Comerota AJ. The ATTRACT trial: rationale for early intervention for iliofemoral DVT. Perspect Vasc Surg Endovasc Ther. 2009 Dec;21(4):221-4; quiz 224-5. doi: 10.1177/1531003509359311. Epub 2010 Jan 3. PMID 20047905
- See also: Deep Vein Thrombosis — http://www.patient.co.uk/showdoc/23068982

RESULTS

PARTICIPANT FLOW:
Groups:
- A-Intervention: Pharmacomechanical catheter-directed thrombolysis (PCDT) with intrathrombus delivery of rt-PA (maximum allowable total dose 35 mg) into the DVT over a period of up to 24 hours. Three methods of initial rt-PA delivery will be used: 1) Trellis-8 Peripheral Infusion System - maximum first-session rt-PA dose 25 mg; 2) AngioJet Rheolytic Thrombectomy System - maximum first-session rt-PA dose 25 mg; or 3) Catheter-directed rt-PA infusion for up to 24 hours at 0.01 mg/kg/hr (maximum 1.0 mg/hr) via a multisidehole infusion catheter. Before and after PCDT, patients will receive standard DVT therapy as in the Control Arm
  Recombinant tissue plasminogen activator (rt-PA): Pharmacomechanical catheter-directed thrombolysis, consisting of intrathrombus administration of rt-PA using a catheter/device.
- B-Control: Initial anticoagulant therapy with unfractionated heparin, enoxaparin, dalteparin, or tinzaparin, for at least 5 days, overlapped with long-term oral warfarin (target international normalized ratio [INR} 2.0 - 3.0). Elastic compression stockings will be prescribed
Period: Overall Study
Arm/Group | A-Intervention | B-Control
Started | 337 | 355
Completed | 257 | 243
Not Completed | 80 | 112

BASELINE CHARACTERISTICS:
Population: One patient was found not to meet the study inclusion criterion, and was excluded from all analyses by the adjudication committee.
Groups:
- A-Intervention: PCDT with intrathrombus delivery of rt-PA (maximum allowable total dose 35 mg) into the DVT over a period of up to 24 hours. Three methods of initial rt-PA delivery will be used: 1) Trellis-8 Peripheral Infusion System - maximum first-session rt-PA dose 25 mg; 2) AngioJet Rheolytic Thrombectomy System - maximum first-session rt-PA dose 25 mg; or 3) Catheter-directed rt-PA infusion for up to 24 hours at 0.01 mg/kg/hr (maximum 1.0 mg/hr) via a multisidehole infusion catheter. Before and after PCDT, patients will receive standard DVT therapy as in the Control Arm
  Recombinant tissue plasminogen activator (rt-PA): Pharmacomechanical catheter-directed thrombolysis, consisting of intrathrombus administration of rt-PA using a catheter/device.
- B-Control: Initial anticoagulant therapy with unfractionated heparin, enoxaparin, dalteparin, or tinzaparin, for at least 5 days, overlapped with long-term oral warfarin (target INR 2.0 - 3.0). Elastic compression stockings will be prescribed
- Total: Total of all reporting groups
Arm/Group | A-Intervention | B-Control | Total
Number analyzed (Participants) | 336 | 355 | 691
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [41 to 62] | 53 [43 to 62] | 53 [42 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 134 | 265
  Male | 205 | 221 | 426
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 26 | 41
  Not Hispanic or Latino | 310 | 319 | 629
  Unknown or Not Reported | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 61 | 62 | 123
  White | 265 | 276 | 541
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 18
Body-mass index [Median (Inter-Quartile Range); unit: kilograms per square meter] | 31 [27 to 36] | 30 [26 to 35] | 31 [27 to 35]
Symptom severity score [Count of Participants; unit: Participants] — The Villalta scale was used to define baseline symptom severity
  Participants
    None or very mild (0-4) | 57 | 69 | 126
    Mild (5-9) | 115 | 124 | 239
    Moderate (10-14) | 98 | 94 | 192
    Severe (> 14) | 66 | 66 | 132
    Not documented | 0 | 2 | 2
Side of index DVT [Count of Participants; unit: Participants]
  Left leg | 207 | 218 | 425
  Right leg | 129 | 137 | 266
Previous DVT or PE [Count of Participants; unit: Participants] — DVT = deep vein thrombosis; PE = pulmonary embolism
  Participants | 83 | 87 | 170
Previous ipsilateral DVT [Count of Participants; unit: Participants] — DVT = deep vein thrombosis
  Participants | 5 | 14 | 19
DVT extends into iliac or common femoral vein [Count of Participants; unit: Participants] — Patients with DVT extending into the iliac or common femoral vein are termed "iliofemoral DVT" and those whose DVT did not extend that high are termed "femoropopliteal DVT".
  Participants | 195 | 196 | 391
DVT risk factors [Count of Participants; unit: Participants]
  Major surgery | 27 | 34 | 61
  Hospitalization | 26 | 38 | 64
  Plaster cast immobilization | 8 | 9 | 17
  Childbirth | 3 | 5 | 8
  None of the above risk factors | 272 | 269 | 541
Outpatient [Count of Participants; unit: Participants] | 268 | 300 | 568
Time from symptom start to randomization [Median (Inter-Quartile Range); unit: days] | 6 [4 to 10] | 6 [4 to 9] | 6 [4 to 10]
Aspirin use within past 7 days [Count of Participants; unit: Participants] | 68 | 74 | 142
Estimated glomerular filtration rate [Median (Inter-Quartile Range); unit: milliliters per minute] | 86 [70 to 102] | 86 [71 to 102] | 86 [71 to 102]
Hypertension [Count of Participants; unit: Participants] | 143 | 139 | 282
Diabetes [Count of Participants; unit: Participants] | 59 | 54 | 113
High cholesterol [Count of Participants; unit: Participants] | 97 | 105 | 202
Asthma [Count of Participants; unit: Participants] | 36 | 38 | 74
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] — COPD = chronic obstructive pulmonary disease
  Participants | 9 | 15 | 24
Angina or myocardial infarction [Count of Participants; unit: Participants] — MI = myocardial infarction
  Participants | 13 | 15 | 28
Congestive heart failure [Count of Participants; unit: Participants] | 13 | 19 | 32
Height [Mean (Standard Deviation); unit: centimeters] | 174 (11) | 174 (10) | 174 (11)
Weight [Mean (Standard Deviation); unit: kilograms] | 97 (25) | 96 (24) | 97 (24)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Post-Thrombotic Syndrome (Villalta Scale)
Description: Patients who experienced one of the following occurrences in the index leg between the 6 month and 24 month post-randomization follow-up visits, inclusive: 1) Villalta score of 5 or greater; 2) leg ulcer; or 3) late endovascular procedure performed to treat severe venous disease. The Villalta scale ranges from 0-33 points, with higher scores being worse.
Time Frame: Between 6 and 24 months after randomization
Population: Modified full analysis set; intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 157 | 171
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.56, Cochran-Mantel-Haenszel; Adjusted for extent of DVT and for clinical center; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.82 to 1.11] — Numerator: PCDT Arm; Denominator: Control Arm. Primary outcome = no statistically significant difference between the two arms

2. Secondary Outcome: Major Non-post-thrombotic Syndrome Treatment Failure
Description: A major non-post-thrombotic-syndrome treatment failure refers to when any of three events occurred in the index leg: 1) an unplanned endovascular procedure to treat severe venous symptoms within 6 months post-randomization; 2) venous gangrene within 6 months; or 3) an amputation within 24 months.
Time Frame: Through 24 months
Population: Modified full analysis set; intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 4 | 7
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.38, Cochran-Mantel-Haenszel; Adjusted by extent of thrombus and clinical center; Risk Ratio (RR) = 0.58, 95% CI 2-sided [0.17 to 1.98] — Numerator: PCDT Arm; Denominator: Control Arm. No statistically significant difference was seen

3. Secondary Outcome: Any Treatment Failure
Description: Composite of PTS and major non-PTS treatment failure
Time Frame: Through 24 months
Population: Modified full analysis set; intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 158 | 176
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.39, Cochran-Mantel-Haenszel; Adjusted for thrombus extent and clinical center; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.80 to 1.09] — No statistically significant difference was seen

4. Secondary Outcome: Moderate-to-severe Post-thrombotic Syndrome
Description: Proportion of patients with Villalta score of 10 or higher at any time between the 6 month and 24 month follow-up visits, inclusive. The Villalta scale ranges from 0-33 points, with higher scores being worse.
Time Frame: Between 6 and 24 months after randomization
Population: Modified full analysis set, intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 60 | 84
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.04, Cochran-Mantel-Haenszel; Adjusted by extent of DVT and clinical center; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.54 to 0.98] — Numerator: PCDT Arm; Denominator: Control Arm

5. Secondary Outcome: Major Bleeding
Description: Defined as clinically overt bleeding that is associated with a fall in the hemoglobin level of at least 2.0 g/dl, transfusion of ≥ 2 units of red blood cells, or involvement of a critical site (e.g. intracranial, intraspinal).
Time Frame: Within 10 days after randomization
Population: Modified full analysis set, intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 6 | 1
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.049, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 6.18, 95% CI 2-sided [0.78 to 49.2] — Numerator: PCDT Arm; Denominator: Control Arm. More major bleeding was observed in the PCDT Arm

6. Secondary Outcome: Major Bleeding
Description: Defined as clinically overt bleeding that was associated with a fall in the hemoglobin level of at least 2.0 g/dl, transfusion of ≥ 2 units of red blood cells, or involvement of a critical site (e.g. intracranial, intraspinal).
Time Frame: Within 24 months after randomization
Population: Modified full analysis set; intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 19 | 13
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.23, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.52, 95% CI 2-sided [0.76 to 3.01] — Numerator: PCDT Arm; Denominator: Control Arm

7. Secondary Outcome: Any (Minor + Major) Bleeding
Description: Clinically overt bleeding that occurred through 10 days post-randomization
Time Frame: Within 10 days after randomization
Population: Modified full analysis set, intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 15 | 6
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.03, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 2.64, 95% CI 2-sided [1.04 to 6.68] — Numerator = PCDT Arm; Denominator = Control Arm. Bleeding was more frequent in the PCDT Arm

8. Secondary Outcome: Any (Major + Minor) Bleeding
Description: Clinically overt bleeding that occurred within 24 months post-randomization
Time Frame: Within 24 months after randomization
Population: Modified full analysis set, intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 46 | 38
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.25, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.26, 95% CI 2-sided [0.85 to 1.89] — Numerator: PCDT Arm; Denominator: Control Arm

9. Secondary Outcome: Recurrent Venous Thromboembolism
Description: Proportion of patients with symptomatic recurrent venous thromboembolism (including DVT and/or PE)
Time Frame: Within 10 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 6 | 4
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.50, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.53, 95% CI 2-sided [0.44 to 5.28] — Numerator = PCDT Arm; Denominator = Control Arm

10. Secondary Outcome: Recurrent Venous Thromboembolism
Description: Symptomatic recurrent venous thromboembolism (DVT and/or PE)
Time Frame: Within 24 months after randomization
Population: Modified full analysis set; intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 42 | 30
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.09, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.47, 95% CI 2-sided [0.94 to 2.29] — Numerator: PCDT Arm; Denominator: Control Arm

11. Secondary Outcome: Death
Description: All-cause mortality
Time Frame: Within 10 days after randomization
Population: Modified full analysis set; intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 0 | 0

12. Secondary Outcome: Death
Description: All-cause mortality
Time Frame: Within 24 months after randomization
Population: Modified full analysis set; intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 336 | 355
Participants | 7 | 8
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.83, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.33 to 2.44]

13. Secondary Outcome: Severity of Post-thrombotic Syndrome (Villalta)
Description: Mean Villalta scale score at the specified follow-up visit. Villalta score ranges from 0-33 points, with higher scores being worse.
Time Frame: At 6 months
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 291 | 285
points | 3.11 (0.24) | 4.33 (0.24)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p < 0.001, Regression, Linear; Piecewise linear-regression growth-curve models with adjustment for extent of DVT, clinical center) and pre-specified baseline co-variates; Mean Difference (Net) = -1.22, Standard Error of Mean 0.31 — Lower (better) mean scores in the PCDT Arm

14. Secondary Outcome: Severity of Post-thrombotic Syndrome (Villalta)
Description: as for outcome 13
Time Frame: At 12 months
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 272 | 258
points | 3.22 (0.22) | 4.38 (0.22)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p < 0.001, Regression, Linear; [statistical method as in outcome 13, analysis 1]; Mean Difference (Net) = -1.17, Standard Error of Mean 0.28 — Lower (better) mean scores in the PCDT Arm

15. Secondary Outcome: Severity of Post-thrombotic Syndrome (Villalta)
Description: Mean Villalta scale score at specified follow-up visit. Villalta score ranges from 0-33 points, with higher scores being worse.
Time Frame: At 18 months
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 245 | 222
points | 3.32 (0.24) | 4.44 (0.24)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p < 0.001, Regression, Linear; [statistical method as in outcome 13, analysis 1]; Mean Difference (Net) = -1.12, Standard Error of Mean 0.31 — Lower (better) mean scores in the PCDT Arm

16. Secondary Outcome: Severity of Post-thrombotic Syndrome (Villalta)
Description: as for outcome 15
Time Frame: At 24 months
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 258 | 239
points | 3.43 (0.28) | 4.50 (0.29)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.005, Regression, Linear; [statistical method as in outcome 13, analysis 1]; Mean Difference (Net) = -1.06, Standard Error of Mean 0.38 — Lower (better) mean scores in the PCDT Arm

17. Secondary Outcome: Venous Clinical Severity Score
Description: Mean Venous Clinical Severity Score (VCSS) at the specified follow-up visit; range 0-27 (did not use compression item), higher score is worse
Time Frame: At 6 months
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 289 | 279
points | 1.73 (0.15) | 2.68 (0.15)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p < 0.001, Regression, Linear; [statistical method as in outcome 13, analysis 1]; Mean Difference (Net) = -0.95, Standard Error of Mean 0.21 — Lower (better) mean scores in the PCDT Arm

18. Secondary Outcome: Venous Clinical Severity Score
Description: Mean VCSS score at the specified follow-up visit; range 0-27 (did not use compression item)
Time Frame: At 12 months
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 265 | 253
points | 1.80 (0.16) | 2.37 (0.16)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.01, Regression, Linear; [statistical method as in outcome 13, analysis 1]; Mean Difference (Net) = -0.56, Standard Error of Mean 0.23 — Lower (better) mean scores in the PCDT Arm

19. Secondary Outcome: Venous Clinical Severity Score
Description: Mean VCSS score at the specified follow-up visit; range 0-27 (did not use compression item)
Time Frame: At 18 months
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 240 | 215
points | 1.74 (0.17) | 2.80 (0.18)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p < 0.001, Regression, Linear; [statistical method as in outcome 13, analysis 1]; Mean Difference (Net) = -1.06, Standard Error of Mean 0.24 — Lower (better) mean scores in the PCDT Arm

20. Secondary Outcome: Venous Clinical Severity Score
Description: Mean VCSS score at the specified follow-up visit; range 0-27 (did not use compression item)
Time Frame: At 24 months
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 235 | 214
points | 1.87 (0.18) | 2.42 (0.19)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.03, Regression, Linear; [statistical method as in outcome 13, analysis 1]; Mean Difference (Net) = -0.55, Standard Error of Mean 0.26 — Lower (better) mean scores in the PCDT Arm

21. Secondary Outcome: Change in General Quality of Life - Physical
Description: Short-Form-36 Health Survey, Version 2, Physical Component Summary (PCS) Scale. Range of scores 0-100 with higher scores representing better quality of life.
Time Frame: Baseline to 24 months post-randomization
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 245 | 222
units on a scale | 11.18 (0.91) | 10.06 (2.70)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.37, Regression, Linear; Adjusted by extent of thrombus and clinical center; Mean Difference (Net) = 1.13, Standard Error of Mean 1.26 — No significant difference was seen in the degree of change from baseline to 24 months between the two treatment arms

22. Secondary Outcome: Change in General Quality of Life - Mental
Description: Short-Form-36 Health Survey, Version 2, Mental Component Summary (MCS) Scale. Range of scores 0-100 with higher scores representing better quality of life.
Time Frame: Baseline to 24 months post-randomization
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 245 | 222
units on a scale | 2.70 (0.84) | 2.70 (0.89)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.99, Regression, Linear; Adjusted by extent of thrombus and clinical center; Mean Difference (Net) = 0.00, Standard Error of Mean 1.16 — No difference was observed in the degree of change from baseline to 24 months in the two treatment groups

23. Secondary Outcome: Change in Venous Disease-specific Quality of Life
Description: Venous Insufficiency Epidemiological and Economic Study Quality of Life (VEINES-QOL) questionnaire. Range of scores 0-100 with higher scores representing better quality of life, and higher change scores representing greater improvement from baseline.
Time Frame: Baseline to 24 months post-randomization
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 249 | 226
units on a scale | 27.67 (1.71) | 23.47 (17.31)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.08, Regression, Linear; Adjusted by extent of thrombus and clinical center; Mean Difference (Net) = 4.20, Standard Error of Mean 2.39 — No significant difference in the change from baseline to 24 months between the two treatment arms

24. Secondary Outcome: Change in Leg Pain Severity
Description: Likert pain scale ranging from 1-7, with higher scores representing a greater intensity of pain
Time Frame: Baseline to 10 days post-randomization
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 317 | 325
points | -1.62 (0.10) | -1.29 (0.10)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.02, Regression, Linear; Adjusted by extent of thrombus and clinical center; Mean Difference (Net) = -0.33, Standard Error of Mean 0.14

25. Secondary Outcome: Change in Leg Pain Severity
Description: Likert pain scale ranging from 1-7, with higher scores representing a greater intensity of pain
Time Frame: Baseline to 30 days post-randomization
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: points
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 314 | 317
points | -2.17 (0.11) | -1.83 (0.11)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.03, Regression, Linear; Adjusted by extent of thrombus and clinical center; Mean Difference (Net) = -0.34, Standard Error of Mean 0.15

26. Secondary Outcome: Change in Leg Circumference
Description: Mean calf circumference measured 10 cm below the tibial tuberosity
Time Frame: Baseline to 10 days post-randomization
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 305 | 323
centimeters | -0.26 (0.17) | 0.27 (0.16)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.02, Regression, Linear; Adjusted by extent of thrombus and clinical center; Mean Difference (Net) = -0.53, Standard Error of Mean 0.23

27. Secondary Outcome: Change in Leg Circumference
Description: Mean calf circumference measured 10 cm below the tibial tuberosity
Time Frame: Baseline to 30 days post-randomization
Population: Modified full analysis set; intention to treat
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | A-Intervention | B-Control
Number analyzed (Participants) | 304 | 315
centimeters | -0.74 (0.17) | -0.28 (0.16)
Statistical Analysis 1: Comparison: A-Intervention vs B-Control; Test type: Superiority; p = 0.05, Regression, Linear; Adjusted by extent of thrombus and clinical center; Mean Difference (Net) = -0.46, Standard Error of Mean 0.23

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected throughout the study - i.e. through 24 months post-randomization. Non-serious adverse events were collected through 30 days post-randomization, and through 30 days after any subsequent PCDT procedure.
Arm/Group | A-Intervention | B-Control
All-Cause Mortality (participants affected / at risk) | 7/336 | 8/355
Serious Adverse Events (participants affected / at risk) | 109/336 | 86/355
Other Adverse Events (participants affected / at risk) | 0/336 | 0/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-Intervention (N=336) | B-Control (N=355)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 4 (4)
Abnormal lab results secondary to undetermined infection (Infections and infestations) | 1 (1) | 0 (0)
Acute and progressive cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Acute arterial limb ischemia of left lower extremity (Vascular disorders) | 1 (1) | 0 (0)
Acute CHF with atrial fibrillation and rapid ventricular response (Cardiac disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute diverticulitis (Infections and infestations) | 0 (0) | 1 (2)
Acute encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Acute gallstone pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Acute on chronic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute on chronic respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute oxycodone and doxylamine intoxication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute phencyclidine intoxication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute rejection (heart transplant) (Cardiac disorders) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 5 (7) | 1 (4)
Acute right lower extremity DVT and acute bronchitis (Vascular disorders) | 0 (0) | 1 (1)
Acute short bowel obstruction versus Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute thrombocytopenic purpura (Immune system disorders) | 0 (0) | 1 (1)
Acute viral gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Adenocarcinoma of unknown primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Alcohol intoxication (Injury, poisoning and procedural complications) | 2 (3) | 3 (3)
Alcohol Withdrawal (Psychiatric disorders) | 3 (4) | 0 (0)
Altered mental state (Psychiatric disorders) | 0 (0) | 1 (1)
Anemia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Angioedema, unclear etiology (Immune system disorders) | 1 (3) | 0 (0)
Antral gastritic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aortic insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arterial occlusion (Vascular disorders) | 0 (0) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (19) | 4 (5)
Atrial flutter with rapid ventricular response (Cardiac disorders) | 0 (0) | 1 (1)
Atypical chest pain (Cardiac disorders) | 1 (1) | 2 (2)
Back spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1) | 1 (1)
Bilateral lower extremity cellulitis and CHF (Infections and infestations) | 0 (0) | 1 (1)
Biliary diskinesia and sludge (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bleeding at sheath puncture site (Vascular disorders) | 1 (1) | 0 (0)
Bleeding from wound (Vascular disorders) | 0 (0) | 1 (1)
Bleeding gums (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blurred vision and diffuse itching (Nervous system disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast intraductal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Broken ribs (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
C5 on C6 retrolisthesia (Nervous system disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 6 (7) | 4 (4)
Chest pain (General disorders) | 7 (7) | 10 (11)
Chest pain/asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chest pain and shortness of breath (Cardiac disorders) | 0 (0) | 3 (3)
Chest pain, shortness of breath, hemoptysis (Cardiac disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (8)
Colitis (Gastrointestinal disorders) | 1 (3) | 1 (1)
Colon cancer - adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Complex gouty septic olecranon bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Congestive heart failure (Cardiac disorders) | 4 (4) | 2 (6)
Coronary artery disease (Cardiac disorders) | 3 (3) | 0 (0)
Coronary artery disease and hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Death secondary to metastatic gastric carcinoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Debridement of right below-the-knee amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Degenerative joint disease with total right hip replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Disconnected VP shunt (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diverticulosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
DVT and PE (Vascular disorders) | 3 (3) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea with lower extremity edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Elevated INR (Investigations) | 1 (1) | 2 (2)
Elevated troponin (Investigations) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Esophageal stricture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall after alcohol abuse (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Foot pain/burning (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fracture and cellulitis of right first toe (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured humerus and ribs - fell off ladder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gangrene left hallux (Infections and infestations) | 1 (1) | 0 (0)
Gastric adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 8 (8) | 6 (6)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gunshot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Hemoperitoneum of unknown etiology (Vascular disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemorrhagic cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhagic shock (Vascular disorders) | 1 (1) | 0 (0)
Heparin induced thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Herniated lumbar disc (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive urgency with CHF exacerbation (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolemic shocck (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia due to hypoventilation due to multiple pain medications (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Influenza A (Infections and infestations) | 0 (0) | 1 (1)
Intertigo labialis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal fluid collection secondary to bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intra-abdominal infection (Infections and infestations) | 1 (2) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Kidney cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lactic acidosis, acute sepsis, atrial fibrillation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Left C4-C5 neuroforaminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left hip removal of hardware and total hip arthoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Left lower extremity pain and abscess (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Leg pain and swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Leg swelling (Cardiac disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lightheadedness (Cardiac disorders) | 1 (1) | 0 (0)
Low hemoglobin (Investigations) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Mania, bizarre behavior, agitation (Investigations) | 0 (0) | 1 (1)
Massive closed head injury (Nervous system disorders) | 1 (1) | 0 (0)
Mediastinal adenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Metastatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Migrated VP shunt (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Methicillin-resistant Staphylococcus Aureus - wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multisystem organ failure (General disorders) | 1 (1) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea, vomiting, diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Non-ST wave myocardial infarction (Cardiac disorders) | 3 (5) | 0 (0)
Obstipation with ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructing ureteral stone (Renal and urinary disorders) | 0 (0) | 1 (1)
Orthostatic hyptension secondary to beta blockers and dehydration (Vascular disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Perihepatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Peripheral arterial disease (Vascular disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleuritic chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (5) | 6 (6)
Pneumonia and pulmonary hypertension likely due to PE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Post-operative infection (Infections and infestations) | 0 (0) | 1 (1)
Post-percardiotomy syndrome (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 7 (9)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 25 (36) | 17 (20)
Renal vein obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Reversible cerebral vasoconstriction syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Right foot amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Right hand abscess (Infections and infestations) | 0 (0) | 1 (1)
Right knee hematoma (Vascular disorders) | 0 (0) | 1 (1)
Right knee tear of medial meniscus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ruptured ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 5 (6)
Sepsis and pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 2 (2)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0)
Severe bilateral knee degenerative joint disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Short-term memory impairment of uncertain etiology (Psychiatric disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Spinal headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Squamous cell carcinoma of unknown primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Staph infection in right shoulder (Infections and infestations) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 6 (6) | 0 (0)
Subdural hematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (6)
Suicidal ideation and alcohol withdrawal (Psychiatric disorders) | 0 (0) | 1 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Surgical excision of squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Suspected infection to stump from right below-knee amputation (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 5 (6)
Syncope and head contusion (Vascular disorders) | 0 (0) | 1 (1)
Transient dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischemia attack (Nervous system disorders) | 0 (0) | 1 (1)
Type A ascending aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract infection and cellulitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Uterine cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ventricular perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Viral gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Viral syndrome (Infections and infestations) | 0 (0) | 1 (1)
Vomoting and diarrhea (Infections and infestations) | 0 (0) | 1 (1)
Venous thromboembolism (Vascular disorders) | 0 (0) | 1 (1)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0)
Retroperitoneal bleed (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes